CLINICAL TRIAL: NCT05517642
Title: Immunogenicity, Efficacy and Safety of Inhaled (IH) Viral Vectored Vaccine (Convidecia, CanSino) as Second Booster Dose Against Emerging Variants of Concern (VOC) of SARS-CoV-2 to Prevent Breakthrough Infections. A Randomized Observer-blind Controlled Trial.
Brief Title: IH Convidecia as Second Booster Dose Against Breakthrough Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CT 2022-01
Record Dates: First submitted 2022-08-22; First posted 2022-08-26 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: Inhaled; Convidecia; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a ratio of 1:1 to receive a second booster dose of IH Convidecia vaccine (treatment arm), or a second booster dose of mRNA vaccine BNT162b2 (Pfizer).
Who Masked: Investigator
Masking Description: Observer-blind clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ad5-nCoV-IH (Experimental): Participates age 18 or older who have completed a course of primary and first booster vaccination at least 16 weeks before, and who have sub-optimal antibody response to the first booster dose, will receive a second booster dose of IH Convidecia vaccine.
  Interventions: Biological: Recombinant COVID-19 vaccine (adenovirus type 5 vector) for Inhalation (Ad5-nCoV-IH)
- mRNA vaccine BNT162b2 (Pfizer) (Active Comparator): Participates age 18 or older who have completed a course of primary and first booster vaccination at least 16 weeks before, and who have sub-optimal antibody response to the first booster dose,will receive a second booster dose of mRNA vaccine BNT162b2 (Pfizer).
  Interventions: Biological: mRNA vaccine BNT162b2 (Pfizer)

INTERVENTIONS:
Biological: Recombinant COVID-19 vaccine (adenovirus type 5 vector) for Inhalation (Ad5-nCoV-IH) — Subjects will be randomized to receive a second booster dose of IH Convidecia vaccine (treatment arm)
  Arms: Ad5-nCoV-IH
Biological: mRNA vaccine BNT162b2 (Pfizer) — Subjects will be randomized to receive a second booster dose of BNT162b2.
  Arms: mRNA vaccine BNT162b2 (Pfizer)

SUMMARY:
This will be a randomized single-blind controlled trial to determine the immunogenicity, efficacy and safety of IH Convidecia (CanSino), as a second booster vaccination against Omicron and other emerging VOCs to prevent breakthrough infections among people with a sub-optimal immune response to the first booster dose.

These subjects will be randomized in a ratio of 1:1 to receive a second booster dose of IH Convidecia vaccine (treatment arm), or a second booster dose of mRNA vaccine BNT162b2 (Pfizer).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give written informed consent for participation in the study.
* Male or Female, aged 18 years or above and in good health as determined by study clinician. Participants may have well controlled or mild-moderate comorbidity.
* Female participants of childbearing potential must be willing to ensure that they or their partner use effective contraception from 1 month prior to first immunisation continuously until 3 months after boost immunisation.
* In the Investigator's opinion, participant is able and willing to comply with all trial requirements.
* At least 16 weeks after first booster dose of vaccination.

Exclusion Criteria:

* Confirmed cases, suspected cases or asymptomatic cases of COVID-19.
* Self-reported history of SARS and MERS infection.
* Receipt of live attenuated vaccine within one month prior to vaccination and other vaccines within 14 days prior to vaccination.
* Receipt of any SARS-COV-2 vaccine after first dose of booster vaccination.
* Participants who are pregnant at enrolment or planning to become pregnant during the first 3 months following vaccination.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of study vaccines.
* Any history of anaphylaxis.
* Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or continuous use of anticoagulants (warfarin, apixaban, rivaroxaban, dabigatran, edoxaban), or prior history of significant bleeding or bruising following IM injections or venipuncture.
* Suspected or known current alcohol or drug dependency.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness (mild/moderate well controlled comorbidities are allowed).
* Participant with life expectancy of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Level of saliva IgA antibodies by ELISA. | 28 days post booster vaccination
Level of serum functional neutralizing antibodies by cPass Genscript | 28 days post booster vaccination
Level of serum Anti-Spike IgG by ELISA. | 28 days post booster vaccination
Level of anti S-RBD IgG by ELISA. | 28 days post booster vaccination
Level of serum Anti-Nucleocapsid IgG by ELISA. | 28 days post booster vaccination
Baseline level of Anti-Ad5 antibodies by ChemiLuminescence. | Day 0
Level of pseudo neutralising antibodies against the wild-type original strain and Beta, Delta, Omicron and emerging VOCs by ELISA. | 28 days post booster vaccination

SECONDARY OUTCOMES:
Incidence of solicited adverse events | 14 days
  Incidence of solicited adverse events post booster vaccination in all subjects.
Incidence of serious adverse events | Up to 24 weeks
  Incidence of serious adverse events post booster vaccination in all subjects.
Incidence of adverse events of special interest (AESI) | Up to 24 weeks
  Incidence of AESI post booster vaccination in all subjects.
Efficacy against COVID-19 infection and transmission | At least 14 days post booster dose.
  RT-PCR-confirmed Covid-19 breakthrough infection, whether symptomatic or not.
Efficacy against COVID-19 infection and transmission | Within 7 days after the sample date of the index case.
  RT-PCR-confirmed Covid-19 secondary attack rate among household members after an index case is detected.
Level of saliva IgA antibodies by ELISA. | 14 days post booster vaccination
Level of serum functional neutralizing antibodies by cPass Genscript | 14 days post booster vaccination
Level of serum Anti-Spike IgG by ELISA. | 14 days post booster vaccination
Level of anti S-RBD IgG by ELISA. | 14 days post booster vaccination
Level of T cell responses by Intracellular Cytokine Staining (Th1/Th2) in subgroup subjects. | Up to 24 weeks
Level of T cell response by Enzyme-linked Immunospot (Elispot) in subgroup subjects. | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Shi Min Ng, Principal Investigator — Hospital Ampang; Norliza Zainudin, Principal Investigator — Hospital Selayang; Sunita Bavanandam, Principal Investigator — Kuala Lumpur General Hospital
Locations (1):
- Hospital Ampang, Ampang, Selangor, Malaysia

REFERENCES:
- [Derived] Chew CK, Wang R, Bavanandan S, Zainudin N, Zhao X, Ahmed S, Nair D, Hou L, Yahya R, Ch'ng SS, Pang LH, Abdul Aziz A, Huang H, Rajasuriar R, Wu S, Zhang Z, Wang X, Chun GY, Mohd Norzi A, Cheah KY, Lee YL, Wan Mohamad WH, Mohd Din MR, Wan Ahmad Kamil WMR, Tan MH, Xu X, Wang L, Yan M, Liu Y, Chin VK, Teo JS, Lim TO, Zhu T, Gou J, Ng SSM. Safety, efficacy and immunogenicity of aerosolized Ad5-nCoV COVID-19 vaccine in a non-inferiority randomized controlled trial. NPJ Vaccines. 2024 Oct 31;9(1):209. doi: 10.1038/s41541-024-01003-x. PMID 39482336